CLINICAL TRIAL: NCT07235358
Title: Glycemic Effects of Substituting Pecans for Snacks Higher in Saturated Fat and Added Sugars in Individuals With Prediabetes
Brief Title: Cardiometabolic Effects of Pecan Snacking in Prediabetes
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Penn State University (Other)
Collaborators: American Pecan Promotion Board (Unknown)
Responsible Party: Principal Investigator, Kristina Petersen PhD, APD, FAHA, Associate Professor, Penn State University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: PEC
Record Dates: First submitted 2025-11-14; First posted 2025-11-19 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Prediabetes
Keywords: diet; nutrition; nuts; snacking; prediabetes; cardiovascular disease
MeSH Terms: conditions — Prediabetic State; Cardiovascular Diseases

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pecan snacking group (Experimental): Participants will be provided with 1.5 oz/day of pecans and asked to eat these instead of typically consumed snacks higher in saturated fat and added sugars.
  Interventions: Behavioral: Pecan snacking
- Usual diet (Active Comparator): Participants will be asked to continue consuming their usual diet. To match attention and resources, participants will be provided with a grocery voucher in approximately equivalent value to the pecans.
  Interventions: Other: Usual diet

INTERVENTIONS:
Behavioral: Pecan snacking — Replacement of typically consumed snacks with 1.5 oz/day of pecans
  Arms: Pecan snacking group
Other: Usual diet — Continue with usual diet
  Arms: Usual diet

SUMMARY:
The purpose of this study is to investigate the effects of replacing snacks higher in saturated fats and added sugars with pecans on blood sugar control, heart health and diet quality in individuals with prediabetes. Participants will be randomized into one of two groups. Group 1 will consume 1.5 oz of pecans per day in place of normally consumed snacks higher in saturated fat and added sugars for 16 weeks. Group 2 will be asked to continue consuming their current diet for 16 weeks. Measures will be taken to evaluate blood sugar, heart health and dietary intake at the beginning and 16 weeks later.

DETAILED DESCRIPTION:
This is a 16-week randomized controlled trial. Participants will be randomized to either: 1) replace current snacks higher in saturated fat and added sugars with 1.5 oz/day of pecans; 2) continue their habitual diet. At the beginning and the end of the 16-week study period, testing will be conducted.

ELIGIBILITY:
Inclusion Criteria:

* Age 25-65 years
* Prediabetes assessed by an HbA1c of 5.7-6.4% at screening
* BMI 25-40 kg/m2 at screening
* Low habitual nut consumption (<3.5 oz-eq/week) assessed at the telephone screening
* Regularly eats snacks higher in saturated fat and/or added sugars assessed at the telephone screening

Exclusion Criteria:

* LDL-C ≥190 mg/dL at screening
* Hemoglobin <13.2 g/dL at screening
* Fasting triglycerides >350 mg/dL at screening
* ≥10% change in body weight within the 6 months prior to enrollment
* Blood pressure >140/90 mmHg at screening
* Type 1 or type 2 diabetes
* Prescription of anti-hypertensive, lipid-lowering, or glucose-lowering drugs
* Intake of supplements or over-the-counter medications that affect the outcomes of interest (i.e., lipid, blood pressure, or glucose lowering; vitamin C or multi-vitamins containing vitamin C) and are unwilling to cease during the study period.
* History of liver, kidney, or autoimmune disease
* Prior cardiovascular event (e.g., stroke, heart attack)
* Current pregnancy or intention of pregnancy within the next 12 months
* Lactation within the prior 6 months
* Pecan allergy/intolerance/sensitivity/dislike
* Unwilling/unable to eat 1.5 oz of pecans every day as a snack during the duration of the study
* Antibiotic use within the prior 4 weeks
* Oral steroid use within the prior 4 weeks
* Use of tobacco or nicotine-containing products within the past 6 months
* History of cancer at any site within the past 10 years (eligible if ≥10 years without recurrence) or non-melanoma skin cancer within the past 5 years (eligible if ≥5 years without recurrence)
* Participation in another clinical trial within 60 days of baseline
* Unwilling to contact study staff before enrolling in other health-related research and avoid participating in any research that may interfere with this study.
* Currently following a restricted or weight-loss diet
* Prior bariatric surgery
* Intake of >14 alcoholic drinks/week and/or not willing to avoid alcohol consumption for 48 hours prior to test visits
* Principal Investigator discretion related to the potential participant's ability to adhere to the study requirements, including being able to come to attend visits
* Does not speak and/or understand English
* Unwilling to refrain from donating blood or plasma during the study
* Weight <110 lb
* If a potential participant takes thyroid medicine, abnormal thyroid stimulated hormone (TSH) concentration (TSH outside of normal range), or change in dose of thyroid medication within the last 6 months

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 147 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2027-09-30 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
Change in HbA1c | 16 weeks
  HbA1c will be assessed at baseline and 16-weeks and expressed as percentage . The change in HbA1c will be calculated by subtracting the baseline value from the 16 week value and expressed as percentage point change.

SECONDARY OUTCOMES:
Change in fasting glucose | 16 weeks
  Change in fasting plasma glucose expressed as mg/dL. Change in glucose will be calculated as the mean of the 16 week measures (i.e., mean of day 1 and day 2 values) minus the mean of the baseline measures (i.e., mean of day 1 and day 2 values).
Change in mean glucose | 16 weeks
  Change in mean glucose assessed by a continuous glucose monitor (CGM) expressed as mg/dL. Change in mean glucose will be calculated as mean glucose assessed from 7 days of CGM wear at 16 weeks minus mean glucose assessed from 7 days of CGM wear at baseline.
Change in mean time in range | 16 weeks
  Change in mean time in range (glucose 70-140 mg/dL) assessed by a continuous glucose monitor (CGM) expressed as minutes per day. Change in mean time in range will be calculated as mean time in range assessed from 7 days of CGM wear at 16 weeks minus mean time in range assessed from 7 days of CGM wear at baseline.
Change in glycemic variability | 16 weeks
  Change in mean glycemic variability assessed by a continuous glucose monitor (CGM) expressed as the coefficient of variability. Change in mean glycemic variability will be calculated as mean glycemic variability assessed from 7 days of CGM wear at 16 weeks minus mean glycemic variability assessed from 7 days of CGM wear at baseline.
Change in fasting insulin | 16 weeks
  Change in fasting serum insulin expressed as micro IU/mL. Change in insulin will be calculated as the mean of the 16 week measures (i.e., mean of day 1 and day 2 values) minus the mean of the baseline measures (i.e., mean of day 1 and day 2 values).
Change in homeostatic model of insulin resistance (HOMA-IR) | 16 weeks
  Homeostatic model of insulin resistance (HOMA-IR) will be calculated from insulin and glucose measured from a fasting blood sample. Calculated as (insulin × glucose) / 22.5. Change in HOMA-IR will be calculated as the mean of the 16 week measures (i.e., mean of day 1 and day 2 values) minus the mean of the baseline measures (i.e., mean of day 1 and day 2 values).
Change in the lipoprotein insulin resistance index | 16 weeks
  The lipoprotein insulin resistance index will be calculated from Nuclear Magnetic Resonance assessed lipoprotein concentrations according to a previously described method: Metab, Syndr. Relat. Disord. 12 (8) (2014) 422-429. Change will be calculated by subtracting the baseline value from the 16 week value.
Change in LDL-Cholesterol | 16 weeks
  Assessed from fasting blood draw expressed in mg/dL. Change in LDL-cholesterol will be calculated as the mean of the 16-week measures (i.e., mean of day 1 and day 2 values) minus the mean of the baseline measures (i.e., mean of day 1 and day 2 values).
Change in apolipoprotein B | 16 weeks
  Assessed from fasting blood draw expressed in mg/dL. Change in apolipoprotein B will be calculated by subtracting the baseline value from the 16 week value.
Change in non-HDL cholesterol | 16 weeks
  Assessed from fasting blood draw expressed in mg/dL. Change in non-HDL cholesterol will be calculated as the mean of the 16-week measures (i.e., mean of day 1 and day 2 values) minus the mean of the baseline measures (i.e., mean of day 1 and day 2 values).
Change in Total Cholesterol | 16 weeks
  Assessed from fasting blood draw expressed in mg/dL. Change in total cholesterol will be calculated as the mean of the 16-week measures (i.e., mean of day 1 and day 2 values) minus the mean of the baseline measures (i.e., mean of day 1 and day 2 values).
Change in HDL-Cholesterol | 16 weeks
  Assessed from fasting blood draw expressed in mg/dL. Change in HDL-cholesterol will be calculated as the mean of the 16-week measures (i.e., mean of day 1 and day 2 values) minus the mean of the baseline measures (i.e., mean of day 1 and day 2 values).
Change in Triglycerides | 16 weeks
  Assessed from fasting blood draw expressed in mg/dL. Change in triglycerides will be calculated as the mean of the 16-week measures (i.e., mean of day 1 and day 2 values) minus the mean of the baseline measures (i.e., mean of day 1 and day 2 values).
Change in C-reactive protein | 16 weeks
  Assessed from fasting blood draw expressed in mg/L. Change in C-reactive protein will be calculated as the mean of the 16-week measures (i.e., mean of day 1 and day 2 values) minus the mean of the baseline measures (i.e., mean of day 1 and day 2 values).
Change in Central Systolic and Diastolic Blood Pressure | 16 weeks
  Central blood pressure measured assessed using a SphymoCor Xcel (Atcor Medical) at baseline & 16 weeks. Change will be calculated by subtracting the baseline value from the end point value.
Change in Peripheral Systolic and Diastolic Blood Pressure | 16 weeks
  Peripheral blood pressure measured assessed using a SphymoCor Xcel (Atcor Medical) at baseline & 16 weeks. Change will be calculated by subtracting the baseline value from the end point value.
Change in Carotid-Femoral Pulse Wave Velocity | 16 weeks
  Measured assessed using a SphymoCor Xcel (Atcor Medical) at baseline & 16 weeks. Change will be calculated by subtracting the baseline value from the end point value.
Change in particle size and number of LDL, HDL, triglyceride rich lipoproteins | 16 weeks
  Measured via Nuclear Magnetic Resonance at baseline and 16 weeks. The change will be calculated by subtracting the baseline value from the 16 week value.
Change in Saturated fat intake | 16 weeks
  Assessed from 24-hour recalls completed prior to baseline and at 16 weeks. Change in saturated fat will be calculated as saturated fat intake at 16 weeks minus baseline saturated fat intake.
Change in added sugar intake | 16 weeks
  Assessed from 24-hour recalls completed prior to baseline and at 16 weeks. Change in added sugar intake will be calculated as added sugar intake at 16 weeks minus baseline added sugar intake.
Change in diet quality | 16 weeks
  Assessed from 24-hour recalls completed prior to baseline and at 16 weeks. Diet quality will be calculated according to the Healthy Eating Index-2020 (HEI). Change in HEI will be calculated as HEI at 16 weeks minus baseline HEI.

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data will be deposited into an open access repository once results from all pre-specified primary and secondary outcomes are published.
Supporting Information: Study Protocol, SAP
Time Frame: The SAP and protocol will be posted on clinicaltrials.gov prior to enrollment commencing.